CLINICAL TRIAL: NCT01009242
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Single Dose Evaluation of the Pharmacokinetics, Pharmacodynamics and Safety of IV and Subcutaneous CDP6038 in Subjects With Rheumatoid Arthritis on a Stable Dose of Methotrexate
Brief Title: To Evaluate the Blood Levels and Safety of IV and Subcutaneous CDP6038 in Subjects With Rheumatoid Arthritis Using Methotrexate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RA0010; 2009-010813-57 (EudraCT Number)
Record Dates: First submitted 2009-11-04; First posted 2009-11-06 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Arthritis; Rheumatoid Arthritis
Keywords: CDP6038
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid | interventions — olokizumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.1mg/kg and 1mg/kg CDP6038 IV and Placebo IV (Experimental): Cohort 1, Group 1 will compare 0.1mg/kg, 1mg/kg CDP6038 and placebo IV.
  Interventions: Biological: CDP6038; Other: Placebo IV; Drug: Methotrexate
- 1 mg/kg CDP6038 SC and Placebo SC (Experimental): Cohort 1, Group 2 will compare 1mg/kg CDP6038 and placebo sc.
  Interventions: Biological: CDP6038; Other: Placebo SC; Drug: Methotrexate
- Optimized CDP6038 SC (Experimental): Cohort 2, Group 3 will compare optimized sc doses of CDP6038 based on outcome of Cohort 1 with placebo.
  Interventions: Drug: CDP 6038 SC; Drug: Methotrexate

INTERVENTIONS:
Biological: CDP6038 — Single dose:
  1 mg/kg CDP6038 IV
  Arms: 0.1mg/kg and 1mg/kg CDP6038 IV and Placebo IV
Biological: CDP6038 — Single dose:
  0.1mg/kg CDP6038 IV
  Arms: 0.1mg/kg and 1mg/kg CDP6038 IV and Placebo IV
Biological: CDP6038 — Single dose:
  1.0mg/kg CDP6038 SC
  Arms: 1 mg/kg CDP6038 SC and Placebo SC
Other: Placebo IV — Single dose:
  Placebo IV
  Arms: 0.1mg/kg and 1mg/kg CDP6038 IV and Placebo IV
Other: Placebo SC — Single dose:
  Placebo SC
  Arms: 1 mg/kg CDP6038 SC and Placebo SC
Drug: CDP 6038 SC — Optimized CDP6038 SC doses based on outcome of Cohort 1 with placebo
  Arms: Optimized CDP6038 SC
Drug: Methotrexate — Individual stable doses of methotrexate.

SUMMARY:
The primary objectives are to determine the relationship between blood levels of CDP6038 and suppression of C-reactive Protein (CRP) following single doses given as intravenous (IV) infusion or subcutaneous (SC) injection to Rheumatoid Arthritis (RA) patients. The safety of CDP6038 will also be evaluated.

DETAILED DESCRIPTION:
The secondary objectives of the study include determination of the absolute bioavailability of CDP6038 given via sc administration compared with iv infusion; assessment of the immunogenicity potential of single dose CDP6038 and assessment, on an exploratory basis, of other relevant systemic biomarkers and changes in clinical response.

ELIGIBILITY:
Inclusion Criteria:

* RA > 6 months duration on stable Methotrexate
* ≤9 swollen and ≤9 tender joints (28 joint count)
* Minimum Screening CRP of 0.5mg/L

Exclusion Criteria:

* Participation in previous studies with defined agents and durations
* Previous treatment with defined agents and durations
* Presence of, or history of defined medical conditions including those particularly associated with deficiency in immune response
* Pregnancy
* Positive tests/signs of possible latent/active tuberculosis
* Positive HIV
* Drug addiction or alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
PK/PD relationship between systemic CDP6038 exposure and CRP suppression. | For 12 weeks following single dose
Evaluate the safety and tolerability of single doses of CDP6038 For 12 weeks following single dose | For 12 weeks following single dose

SECONDARY OUTCOMES:
Absolute bioavailability of CDP6038 given by sc injection in comparison with iv infusion | For 12 weeks following single dose
Assess the immunogenicity of single dose CDP6038 | Multiple sampling from 0 to 12 weeks following single dose
Assess, on an exploratory basis, changes in clinical response and other systemic biomarkers associated with RA | For 12 weeks following single dose

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (6):
- United States (3):
  - Duncansville, Pennsylvania
  - Dallas, Texas
  - San Antonio, Texas
- Germany (3):
  - Berlin
  - Cologne
  - Erlangen